CLINICAL TRIAL: NCT01684176
Title: Pharmacist Intervention Programme to Improve Medication Adherence in Stroke Patients
Brief Title: Tailored Intervention to Improve Patient Adherence to Secondary Stroke Prevention Medication
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Ulla Hedegaard, PhD student, MSc (pharm), Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AKF-381
Record Dates: First submitted 2012-09-10; First posted 2012-09-12 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Stroke; Transient Ischemic Attack
Keywords: Stroke; Ischemic Attack, Transient; Medication adherence; Motivational interviewing; Stroke prevention
MeSH Terms: conditions — Stroke; Ischemic Attack, Transient; Medication Adherence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Complex tailored intervention (Experimental): The intervention consists of 3 elements:
  1. Medication review with recommendations focused on antithrombotics and adherence to guidelines and patient´s adherence to medications.
  2. Discharge consultation with an pharmacist using motivational interviewing techniques.
  3. Follow-up telephone calls one week, two months and six months after discharge.
  Interventions: Behavioral: Complex tailored intervention; Behavioral: Usual care
- Usual care (Placebo Comparator): Usual care
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Complex tailored intervention
  Arms: Complex tailored intervention
Behavioral: Usual care

SUMMARY:
Patient suffering a Transient Ischemic Attack (TIA) or stroke are subsequently at high risk of a new stroke, however, poor adherence to secondary prevention medications occurs frequently within this patient group. The purpose of this study is to evaluate whether a complex tailored pharmacist intervention will lead to increased adherence to secondary stroke prevention medications and less new stroke events when compared to a usual care group. Interventions focus on motivational interviewing, medication review and telephone follow up.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years or older
* Patient admitted or receiving ambulatory treatment for an acute transient ischemic attack or ischemic stroke which has occurred within the previous 30 days.
* The patient or a carer usually dispenses the patient's medications
* Written consent

Exclusion Criteria:

* Cognitive or physical impairment that would preclude comprehension of a conversation
* Terminal illness
* Lives in a care home or an institution
* Receives dose dispensed medicine from a pharmacy
* Medicine is dispensed by a nurse in the patient's home
* Correctional mental health patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2012-08; Primary Completion 2013-02 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Medication Adherence to antiplatelets, anticoagulants and statins measured by proportion of days covered (PDC). | One year from inclusion
For antiplatelets, anticoagulants and statins: Percent of patients that are at least 80% adherent (PDC>0.8) | 1 year from inclusion

SECONDARY OUTCOMES:
Medication Adherence to antihypertensives measured by proportion of days covered (PDC) | One year from inclusion
Percent of patients that are at least 80% adherent (PDC>0.8) to antihypertensives | One year from inclusion
Non-persistence with thromboprophylactic agents ( antiplatelets, anticoagulants, statins and antihypertensives) measured by percent of patients that are not supplied with medication for more than 3 continuous months | One year from inclusion
Accept rate for thromboprophylactic agents measured by percent of patients starting treatment within 0-90 days after discharge. | 3 months from discharge
Composite endpoint: stroke, myocardial infarction or cardiovascular death | One year from inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- Odense University Hospital, Odense C, Denmark

REFERENCES:
- [Background] Hedegaard U, Kjeldsen LJ, Pottegard A, Bak S, Hallas J. Multifaceted intervention including motivational interviewing to support medication adherence after stroke/transient ischemic attack: a randomized trial. Cerebrovasc Dis Extra. 2014 Dec 11;4(3):221-34. doi: 10.1159/000369380. eCollection 2014 Sep-Dec. PMID 25598772